CLINICAL TRIAL: NCT06040164
Title: Molecular Study of Oral Dysbacteriosis in People With Prediabetes and Diabetes
Brief Title: Oral Endocannabinoids in People With Prediabetes and Diabetes
Acronym: SMILE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: SMILE
Record Dates: First submitted 2023-07-19; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-03

CONDITIONS: PreDiabetes; Diabetes Mellitus, Type 2; Obesity; Oral Dysbiosis; Mouth Disease
Keywords: Endocannabinoids; Prediabetes; Diabetes Mellitus Type 2; Obesity; Oral Dysbiosis; Oral Disease; Cannabinoids
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Obesity; Mouth Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples will be collected under resting conditions using the passive drooling method, in 15 mL tubes, every 1 min, for 5 min in the same tube. Along with the saliva samples, trained personnel will collect 9 ml of blood samples, under resting conditions, in ethylenediaminetetraacetic acid (EDTA) tubes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ob/Pre/H: obesity, prediabetes and healthy mouth
  Interventions: Other: Observational study
- Ob/Pre/OCD: obesity, prediabetes and oral cavity disease
  Interventions: Other: Observational study
- Ob/Diab/H: obesity, diabetes and healthy mouth
  Interventions: Other: Observational study
- Ob/Diab/OCD: obesity, diabetes and oral cavity disease
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention will be performed

SUMMARY:
This study evaluates the relationship of endocannabinoids in saliva with inflammation and oral dysbacteriosis present in people with periodontal disease and prediabetes/type 2 diabetes

DETAILED DESCRIPTION:
Diabetes is a disease that affects millions of people worldwide, and the number of cases is expected to continue to increase in the coming years. Type 2 diabetes (T2D) is the most common form of diabetes and is closely related to prediabetes, a condition in which blood glucose levels are high but not high enough to be diagnosed as diabetes. Both prediabetes and T2D increase the risk of cardiovascular disease and are also associated with diseases of the oral cavity, such as dental caries and periodontal disease. The presence of pathogenic bacteria in the mouth has been linked to these diseases. The endocannabinoid system, a signaling system in the body that regulates various biological processes, has been found to play an important role in energy homeostasis and is implicated in obesity, prediabetes, and T2D. This study seeks to investigate the role of endocannabinoids and related lipids in diseases of the oral cavity in the context of prediabetes and T2D. A bidirectional relationship has been observed between periodontitis and T2D, with inflammation playing a central role in both diseases. Although subtle differences in the microbial composition of the mouth have been identified in people with diabetes, the exact mechanisms remain unclear. Our findings could open up a promising line of research on the therapeutic potential of cannabinoid drugs for the treatment of this type of complications in people with prediabetes/T2D.

ELIGIBILITY:
Inclusion Criteria:

* Adults, both sexes (40-65 years)
* With obesity and prediabetes: BMI 30-40 and HbA1c 5.7-6.4
* With obesity and diabetes: BMI 30-40 and previous diagnosis of diabetes

Exclusion Criteria:

* Pregnant women
* Diagnosis of some type of neoplasia or treated with radiotherapy and/or chemotherapy in the last year.
* Ongoing inflammatory diseases (Crohn's disease, ulcerative colitis, arthritis, etc.) and/or anti-inflammatory treatments
* Presence of systemic diseases of vital organs
* Participants in treatment with drugs that could alter salivary flow
* Smokers
* Participants who have not followed the specifications prior to sampling
* Participants who did not sign the informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients to enroll will come from three clinical studies led by our unit: The Pizarra study, an epidemiological study of the Endocrinology and Nutrition unit of the Regional Hospital of Malaga that has provided detailed information on anthropometric and biochemical parameters, eating habits and lifestyle in a cohort of about 1700 subjects; the di@bet.es study, a national epidemiological study carried out on a sample of more than 5,000 people; and the April study, a nutritional intervention study in people with obesity and prediabetes. In addition, the obesity databases of the Endocrinology and Nutrition unit of the Regional Hospital of Malaga will also be used.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 2-arachidonoyl-glycerol (2-AG) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in N-arachidonoylethanolamine (AEA) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in N-palmitoylethanolamine (PEA) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in N-oleoylethanolamine (OEA) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in N-palmitoylethanolamine (DHEA) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in 2-linoleoyl-glycerol (2-LG) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in 2-oleoyl-glycerol (2-OG) levels in saliva and plasma | Basal
  Measured in pmol/ml

SECONDARY OUTCOMES:
Change in interleukin-1β levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in interleukin-6 levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in interleukin-8 levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in interleukin-10 levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in interleukin-17 levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in leptin levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in vascular endothelial growth factor (VEGF) levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in Interferon gamma (IFN)-γ levels in saliva and plasma | Basal
  Measured in pmol/ml
Change in Tumor necrosis factor alpha (TNF)-α levels in saliva and plasma | Basal
  Measured in pmol/ml
Changes in oral bacteriological profile | Basal
  Bacterial 16S rRNA amplicon of the following bacterial strains: Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum, Parvimonas micra, Campylobacter rectus, Eikenella corroe, Veillonella parvula and Actinomyces naeslundii for periodontal disease; and Streptococcus mutans, S. sanguis, S. mitior, S. salivarius and S. milleri for dental caries. Unit of Measurement: Fold-increase over reference genes, delta-delta Ct method.
Changes in Fasting glucose levels | Basal
  Measured in mg/dl
Changes in insulin levels | Basal
  Measured in mUI/mL
Changes from baseline HOMA-IR levels | Basal
  HOMA-IR = [blood insulin (mu/L) × Blood glucose (mmol/L)]/22.5
Changes from baseline HOMA2-IR levels | Basal
  The homeostasis model assessment computational method is used to estimate insulin resistance (HOMA2-IR) from fasting plasma glucose and insulin. The HOMA2-IR is the reciprocal of insulin sensitivity (%S), as a percentage of a normal reference population (normal young adult). A higher score indicates a lower insulin sensitivity.
Changes from baseline HOMA2%S levels | Basal
  Measured in %
Changes from baseline HOMA2%B levels | Basal
  Measured in %
Changes from baseline QUICKY levels | Basal
  QUICKY = 1 / (log(fasting insulin μU/mL) + log(fasting glucose mg/dL))
Changes from baseline HbA1c levels | Basal
  Measured in %
BMI (body mass index) changes | Basal
  Calculated as weight ⁄ height (kg/m2)
Changes in waist circumference | Basal
  Measured in cm
Changes in waist/hip ratio | Basal
  Calculated as waist measurement (cm) divided by hip measurement (cm) (W⁄H)
Changes in waist/height ratio | Basal
  Calculated as waist measurement (cm) divided by height measurement (cm), (W/He)
Changes in blood pressure | Basal
  Measured in mmHg
Changes in triglycerides | Basal
  Measured in mg/dL
Changes in total cholesterol | Basal
  Measured in mg/dL
Changes in HDL cholesterol | Basal
  Measured in mg/dL
Changes in LDL cholesterol | Basal
  Measured in mg/dL
Changes in sialometry | Basal
  Measured in mL/min
Changes in salivary viscosity | Basal
  Measured in poise (1 g·(s·cm)-1)
Changes in salivary pH | Basal
  Logarithm of hydrogen ion concentration
Oral health impact profile | Basal
  The Oral Health Impact Profile will be assessed by using the OHIP-14sp questionnaire, which is one of the most internationally spread indicators of oral health-related quality of life and it is used to measure the impact of oral conditions on quality of life to complement clinical data in cross-sectional and longitudinal studies. The OHIP-14 is a self-filled questionnaire that focuses on seven dimensions of impact (functional limitation, pain, psychological discomfort, physical disability, psychological disability, social disability and handicap) with participants being asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score2), fairly often (score 3) and very often (score 4) using a twelve-months recall period.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Bermúdez-Silva, PhD, Principal Investigator — Hospital Regional Universitario de Málaga - FIMABIS

REFERENCES:
- [Background] IDF Diabetes Atlas 10th edition. Accessed September 29, 2022. www.diabetesatlas.org
- [Background] Aleixandre MA, Miguel M. Síndrome metabólico. Endocrinologia y Nutricion. 2007;54(9). doi:10.1016/S1575-0922(07)71487-0
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Bissett SM, Stone KM, Rapley T, Preshaw PM. An exploratory qualitative interview study about collaboration between medicine and dentistry in relation to diabetes management. BMJ Open. 2013 Feb 14;3(2):e002192. doi: 10.1136/bmjopen-2012-002192. Print 2013. PMID 23418299
- [Background] Tavares RDCR, Ortigara GB, Tatsch KF, Ferreira CM, Boligon J, Moreira CHC. Association between periodontitis and glycated hemoglobin levels in individuals living in rural Southern Brazil. Clin Oral Investig. 2021 Dec;25(12):6901-6907. doi: 10.1007/s00784-021-03980-y. Epub 2021 May 31. PMID 34059955
- [Background] Kriebel K, Hieke C, Muller-Hilke B, Nakata M, Kreikemeyer B. Oral Biofilms from Symbiotic to Pathogenic Interactions and Associated Disease -Connection of Periodontitis and Rheumatic Arthritis by Peptidylarginine Deiminase. Front Microbiol. 2018 Jan 30;9:53. doi: 10.3389/fmicb.2018.00053. eCollection 2018. PMID 29441048
- [Background] Canepari P, Zerman N, Cavalleri G. Lack of correlation between salivary Streptococcus mutans and lactobacilli counts and caries in IDDM children. Minerva Stomatol. 1994 Nov;43(11):501-5. PMID 7739481
- [Background] Estrich CG, Araujo MWB, Lipman RD. Prediabetes and Diabetes Screening in Dental Care Settings: NHANES 2013 to 2016. JDR Clin Trans Res. 2019 Jan;4(1):76-85. doi: 10.1177/2380084418798818. Epub 2018 Sep 6. PMID 30596147
- [Background] Kocher T, Holtfreter B, Petersmann A, Eickholz P, Hoffmann T, Kaner D, Kim TS, Meyle J, Schlagenhauf U, Doering S, Gravemeier M, Prior K, Rathmann W, Harks I, Ehmke B, Koch R. Effect of Periodontal Treatment on HbA1c among Patients with Prediabetes. J Dent Res. 2019 Feb;98(2):171-179. doi: 10.1177/0022034518804185. Epub 2018 Oct 16. PMID 30326764
- [Background] Artur C, Otto-Buczkowska E (2014) Oral Health Problems among Diabetic Patients - Part of Dental Professionals in Diagnostic and Therapy. J Oral Hyg Health 2:167. doi:10.4172/2332-0702.1000167
- [Background] Di Marzo V, Silvestri C. Lifestyle and Metabolic Syndrome: Contribution of the Endocannabinoidome. Nutrients. 2019 Aug 20;11(8):1956. doi: 10.3390/nu11081956. PMID 31434293
- [Background] Gatta-Cherifi B, Cota D. New insights on the role of the endocannabinoid system in the regulation of energy balance. Int J Obes (Lond). 2016 Feb;40(2):210-9. doi: 10.1038/ijo.2015.179. Epub 2015 Sep 16. PMID 26374449
- [Background] Bermudez-Silva FJ, Cardinal P, Cota D. The role of the endocannabinoid system in the neuroendocrine regulation of energy balance. J Psychopharmacol. 2012 Jan;26(1):114-24. doi: 10.1177/0269881111408458. Epub 2011 Aug 8. PMID 21824982
- [Background] Di Marzo V. New approaches and challenges to targeting the endocannabinoid system. Nat Rev Drug Discov. 2018 Sep;17(9):623-639. doi: 10.1038/nrd.2018.115. Epub 2018 Aug 17. PMID 30116049
- [Background] Hillard CJ. Circulating Endocannabinoids: From Whence Do They Come and Where are They Going? Neuropsychopharmacology. 2018 Jan;43(1):155-172. doi: 10.1038/npp.2017.130. Epub 2017 Jun 27. PMID 28653665
- [Background] Fabio Arturo, Iannotti and Fabiana, Piscitelli (November 2018)Endocannabinoidome. In: eLS. John Wiley & Sons, Ltd:Chichester.DOI: 10.1002/9780470015902.a0028301
- [Background] Davis, M.P. (2022). Overview of the Endocannabinoid System and Endocannabinoidome. In: Cannabis and Cannabinoid-Based Medicines in Cancer Care. Springer, Cham. https://doi.org/10.1007/978-3-030-89918-9_1
- [Background] Cani PD, Plovier H, Van Hul M, Geurts L, Delzenne NM, Druart C, Everard A. Endocannabinoids--at the crossroads between the gut microbiota and host metabolism. Nat Rev Endocrinol. 2016 Mar;12(3):133-43. doi: 10.1038/nrendo.2015.211. Epub 2015 Dec 18. PMID 26678807
- [Background] Romero-Zerbo SY, Bermudez-Silva FJ. Cannabinoids, eating behaviour, and energy homeostasis. Drug Test Anal. 2014 Jan-Feb;6(1-2):52-8. doi: 10.1002/dta.1594. Epub 2013 Dec 26. PMID 24375977
- [Background] Lalla E, Papapanou PN. Diabetes mellitus and periodontitis: a tale of two common interrelated diseases. Nat Rev Endocrinol. 2011 Jun 28;7(12):738-48. doi: 10.1038/nrendo.2011.106. PMID 21709707
- [Background] Sanz M, Ceriello A, Buysschaert M, Chapple I, Demmer RT, Graziani F, Herrera D, Jepsen S, Lione L, Madianos P, Mathur M, Montanya E, Shapira L, Tonetti M, Vegh D. Scientific evidence on the links between periodontal diseases and diabetes: Consensus report and guidelines of the joint workshop on periodontal diseases and diabetes by the International Diabetes Federation and the European Federation of Periodontology. J Clin Periodontol. 2018 Feb;45(2):138-149. doi: 10.1111/jcpe.12808. Epub 2017 Dec 26. PMID 29280174
- [Background] Rohani B. Oral manifestations in patients with diabetes mellitus. World J Diabetes. 2019 Sep 15;10(9):485-489. doi: 10.4239/wjd.v10.i9.485. PMID 31558983
- [Background] Thorstensson H, Dahlen G, Hugoson A. Some suspected periodontopathogens and serum antibody response in adult long-duration insulin-dependent diabetics. J Clin Periodontol. 1995 Jun;22(6):449-58. doi: 10.1111/j.1600-051x.1995.tb00176.x. PMID 7560223
- [Background] Takahashi K, Nishimura F, Kurihara M, Iwamoto Y, Takashiba S, Miyata T, Murayama Y. Subgingival microflora and antibody responses against periodontal bacteria of young Japanese patients with type 1 diabetes mellitus. J Int Acad Periodontol. 2001 Oct;3(4):104-11. PMID 12666949
- [Background] Prestifilippo JP, Fernandez-Solari J, de la Cal C, Iribarne M, Suburo AM, Rettori V, McCann SM, Elverdin JC. Inhibition of salivary secretion by activation of cannabinoid receptors. Exp Biol Med (Maywood). 2006 Sep;231(8):1421-9. doi: 10.1177/153537020623100816. PMID 16946411
- [Background] Matias I, Gatta-Cherifi B, Tabarin A, Clark S, Leste-Lasserre T, Marsicano G, Piazza PV, Cota D. Endocannabinoids measurement in human saliva as potential biomarker of obesity. PLoS One. 2012;7(7):e42399. doi: 10.1371/journal.pone.0042399. Epub 2012 Jul 31. PMID 22860123
- [Background] Piscitelli F, Di Marzo V. "Redundancy" of endocannabinoid inactivation: new challenges and opportunities for pain control. ACS Chem Neurosci. 2012 May 16;3(5):356-63. doi: 10.1021/cn300015x. Epub 2012 Feb 27. PMID 22860203
- [Background] Andreis K, Billingsley J, Naimi Shirazi K, Wager-Miller J, Johnson C, Bradshaw H, Straiker A. Cannabinoid CB1 receptors regulate salivation. Sci Rep. 2022 Aug 19;12(1):14182. doi: 10.1038/s41598-022-17987-2. PMID 35986066
- [Background] Oral health. Global Burden of Disease Study 2019. Published 2019. Accessed September 30, 2022. https://www.who.int/news-room/fact-sheets/detail/oral-health
- [Background] Ramfjord SP. The Periodontal Disease Index (PDI). J Periodontol. 1967 Nov-Dec;38(6):Suppl:602-10. doi: 10.1902/jop.1967.38.6.602. No abstract available. PMID 5237683

DOCUMENTS (1):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT06040164/Prot_000.pdf